CLINICAL TRIAL: NCT07277049
Title: Optimisation and Outcome Evaluation of a Just-in-time Adaptive Intervention (JITAI) for Sleep and Circadian Problems: A Micro-randomised Trial and a Randomised Controlled Trial
Brief Title: Optimisation and Evaluation of a Just-in-time Adaptive Intervention (JITAI) for Sleep and Circadian Problems (Phase III)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY037
Record Dates: First submitted 2025-11-26; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Sleep and Circadian Problems
Keywords: Just-in-time Adaptive Intervention (JITAI); sleep and circadian problems; sleep-wake patterns; insomnia; sleep; ecological momentary assessment; mHealth
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimised just-in-time adaptive intervention (GoodShleep+) group (Experimental): Just-in-time adaptive interventions (JITAIs) are defined as interventions that combine two characteristics: just-in-time (intervening in exact moments of need to reduce fatigue and improve adherence) and adaptive (selecting and delivering tailored interventions with the right type and amount in an adaptive manner based on the user's dynamic internal state and environment, typically through ecological momentary assessment and wearables). A comprehensive framework for JITAI design encompasses six key elements, including (1) decision points, (2) tailoring variables, (3) intervention options, and (4) decision rules. These decisions are guided by (5) proximal outcomes and (6) distal outcomes.
  The optimised Goodshleep+, which is based on and modified from the intervention protocol 'Transdiagnostic Intervention for Sleep and Circadian Dysfunction' (TranS-C) will be used. Context-based behavioural strategies will be suggested through push notifications based on specific decision rules.
  Interventions: Behavioral: Optimised just-in-time adaptive intervention (JITAI) based on TranS-C (GoodShleep+)
- Care-As-Usual Group (No Intervention): The participants will not receive the Just-in-time Adaptive Intervention (GoodShleep+) but will have access to usual care based on their needs and preferences, including but not limited to pharmacological interventions, psychological interventions, and complementary and alternative medicine. An intervention tracking log will be used to monitor the care the participants receive during the study period. The CAU group will receive GoodShleep+ after completing all the assessments.
  The team will monitor the participants' weekly sleep and circadian functions using PROMIS- SD/SRI and refer those who have serious suicidal risk to the PA for further assessment and professional mental health services if deemed necessary.

INTERVENTIONS:
Behavioral: Optimised just-in-time adaptive intervention (JITAI) based on TranS-C (GoodShleep+) — The JITAI (GoodShleep) will be adjusted and finalised based on the findings from Phase II (MRT) to transform into the optimised JITAI (GoodShleep+).
  The optimized GoodShleep will be an 8-week, sleep- and circadian-targeted intervention programme. The intervention materials will be presented in text format supplemented with diagrams, video/audio clips, quizzes, and culturally relevant examples. Across the 8 sessions, 4 cross-cutting modules will be introduced, including case formulation, sleep and circadian education, motivational interviewing, and goal setting. In addition, the participants will receive 4 core modules addressing sleep-wake regularity, daytime functioning, correcting beliefs, and maintaining behavioral change. Additionally, five selected optional modules will be delivered based on the participant's sleep-wake features and presentations addressing sleep efficiency, excessive time in bed, delayed/advanced sleep phase, sleep-related worry, and nightmares.
  Arms: Optimised just-in-time adaptive intervention (GoodShleep+) group

SUMMARY:
The JITAI approach holds considerable promise for addressing current challenges in mHealth, including the limitations in supporting real-time monitoring, timely intervention, and poor adherence. However, research on JITAIs in the field of behavioural sleep medicine is still in its infancy. Leveraging existing pilot data, this project will entail a micro-randomised trial (MRT) designed to optimise the JITAI components and a randomised controlled trial (RCT) to examine the efficacy of the optimised JITAI on sleep and circadian functions. Specifically, research has indicated that contextually tailored suggestions are more effective in promoting health behaviors compared to generic messages.This study will include personalised, in-the-moment actionable suggestions based on the Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C) to evaluate their efficacy in contrast to generic messages and no notifications.

The proposed project will have three phases. Phase I will be the technological advancement of the JITAI app, GoodShleep. Based on research findings, additional intervention engagement strategies will be added to improve adherence, including personalisation (i.e., personalised feedback and intervention content), gamification (i.e., goal setting and rewards for a completed mission), and reminders (i.e., push notifications). The refined app will be beta-tested by the research team and five individuals experiencing sleep or circadian problems to ensure the app's functionality and usability. Issues that may arise during Phase I will be resolved prior to commencing Phase II.

Phase II will be an MRT aiming to optimise the advanced GoodShleep alongside wearable devices and ecological momentary assessment (EMA). A total of 77 participants with sleep or circadian problems will participate in the JITAI through the advanced GoodShleep, which will comprise (1) an 8-week, smartphone-based JITAI on TranS-C; (2) EMA prompted by push notifications to detect sleep-wake regularity and mood status; and (3) 24-hour real-time wearables assessing sleep and activity. Participants will be randomly assigned to receive contextually personalised suggestions, generic messages, and no notifications based on our micro-randomised algorithm.

Phase III will involve an RCT to evaluate the optimised JITAI app, GoodShleep+ in both short- (immediately after intervention) and medium-term (12 weeks after intervention). Eighty participants with sleep and circadian problems will be randomised into the optimised JITAI (GoodShleep+) and the care-as-usual (CAU) group in a 1:1 allocation ratio. The JITAI (GoodShleep) will be adjusted and finalised based on the findings from Phase II to transform into the optimised JITAI (GoodShleep+). The GoodShleep+ group will receive an 8-week, smartphone-based GoodShleep+ based on TranS-C. The CAU group will not receive the GoodShleep+ but will have access to usual care based on their needs and preferences. The CAU group will receive GoodShleep+ after completing all the assessments. Major assessments will be conducted at baseline, immediate post-intervention and 12-week follow-up. Participants' sleep conditions will be evaluated using the brief consensus sleep diary and wearables. Activity levels will be measured using wearables at multiple time points. Mood status will be assessed using selected items from PANAS-SF. Participants' weekly sleep and circadian functions will be monitored using Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance (SD) and Sleep-Related Impairment (SRI). Other outcomes will include sleep quality, anxiety and depression symptoms, sleep-related cognitions, overall daytime sleepiness, fatigue, quality of life and functional impairment. Intervention acceptability and intervention adherence will also be assessed.

The current registration is only for Phase III of the current research project.

ELIGIBILITY:
Inclusion criteria:

* Adults aged 18 to 65 years living in Hong Kong
* Chinese language fluency and literacy
* Experiencing ≥1 sleep or circadian problems for 3 months based on the Sleep and Circadian Problems Interview, an adapted version of the Insomnia Interview Schedule (i.e., time needed to fall asleep ≥30 minutes for ≥3 nights per week, wake after sleep onset ≥30 minutes for ≥3 nights per week, <6-hour sleep per night or ≥9-hour sleep per night per 24-hour period for ≥3 nights per week, variability in the sleepweek schedule ≥2.78 hours within a week, and falling asleep after 2:00 AM on ≥3 nights per week)
* One or more PROMIS-Sleep Disturbance (PROMIS-SD) item scores ≥4 after reverse scoring
* Having adequate opportunity and circumstances for sleep to occur
* Installing the JITAI app in an Internet-enabled mobile device (iOS or Android operating system)
* Are willing to provide informed consent and comply with the trial protocol.

Exclusion Criteria:

* Involving in any psychological treatment for sleep disturbances in the past 6 months
* Self-report of a significant untreated severe mental illness (e.g., bipolar disorder, psychotic disorder)
* Presence of medical or cognitive disorder(s), or side effects of medication that contribute significantly to sleep or circadian problems or make participation challenging based on the team's clinical judgement
* Working night shift (>2 nights per week) in the past 3 weeks (i.e., regularly scheduled work from 12AM to 6AM)
* Pregnancy or breastfeeding
* Having a medical or psychiatric condition where sleep restriction is deemed unsuitable due to potential worsening of the condition

Other Criteria:

* Individuals who have sleep apnoea or periodic limb movement disorder commonly experience co-occurring insomnia will be included in the study due to the potential benefits they may derive from TranS-C
* To allow for greater generalisability, this study will not exclude those with mental disorders whose conditions are stable based on the research team's judgement
* If serious suicidal risk (i.e., Patient Health Questionnaire Item 9 score >2) is identified, the participant will be referred to the PA (a clinical psychologist) for further assessment and professional mental health services, if needed
* Medication use and changes will be recorded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-02-29 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Patient-Reported Outcomes Measurement Information System-Sleep Disturbance (PROMIS-SD) | Baseline, immediate post-intervention assessment (Week 9), 12-week post-intervention assessment (Week 20)
  8-item scales to assess sleep and circadian functions and impairments
Change in Patient-Reported Outcomes Measurement Information Sleep-Related Impairment (PROMIS-SRI) | Baseline, immediate post-intervention assessment (Week 9), 12-week post-intervention assessment (Week 20)
  8-item scales to assess sleep and circadian functions and impairments

SECONDARY OUTCOMES:
Change in Pittsburgh Sleep Quality Index (PSQI) | Baseline, immediate post-intervention assessment (Week 9), 12-week post-intervention assessment (Week 20)
  A 19-item scale assessing sleep quality over the past month
Change in 7-day Consensus Sleep Diary | 20-week daily survey
  Records sleep time, wake time, perceived sleeping quality, and use of hypnotics on a daily basis
Change in Hospital Anxiety and Depression Scale (HADS) | Baseline, immediate post-intervention assessment (Week 9), 12-week post-intervention assessment (Week 20)
  A 14-item scale measuring anxiety and depression in both hospital and community settings
Change in 16-item version of the Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS-16) | Baseline, immediate post-intervention assessment (Week 9), 12-week post-intervention assessment (Week 20)
  A 16-item scale to assess sleep-related cognitions
Change in Epworth Sleepiness Scale (ESS) | Baseline, immediate post-intervention assessment (Week 9), 12-week post-intervention assessment (Week 20)
  An 8-item scale designed to evaluate overall daytime sleepiness
Change in Multidimensional Fatigue Inventory (MFI) | Baseline, immediate post-intervention assessment (Week 9), 12-week post-intervention assessment (Week 20)
  A 20-item instrument designed to measure fatigue symptoms
Change in Short Form (6-Dimension) Health Survey (SF-6D) | Baseline, immediate post-intervention assessment (Week 9), 12-week post-intervention assessment (Week 20)
  a preference-based single-index measure of the quality of life
Change in Sheehan Disability Scale (SDS) | Baseline, immediate post-intervention assessment (Week 9), 12-week post-intervention assessment (Week 20)
  A 5-item scale to assess functional impairment in work/school, social life and family life
Change in Treatment Acceptability/Adherence Scale (TAAS) | Baseline, immediate post-intervention assessment (Week 9)
  a 10-item scale of the willingness to utilise or recommend the intervention
Change in Credibility-Expectancy Questionnaire (CEQ) | Baseline, immediate post-intervention assessment (Week 9)
  A 6-item scale used to yield ratings of intervention credibility and the expectation of success
Change in System Usability Scale (SUS) | Immediate post-intervention assessment (Week 9)
  A 10-item scale evaluating the usability perception of an app
Change in wearable-derived rest-activity data | 8-week on a daily basis, 24 hours a day
  24-hour rest-activity data will be collected using research-grade wearables (actigraphy). Participants will be instructed to wear the device on their non-dominant wrist, 24 hours a day, for 8 consecutive weeks, with expections during water sports activities.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong